CLINICAL TRIAL: NCT02678884
Title: A Pilot Study of 18F-FDG PET-CT Kinetic Analysis in Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Head and Neck Squamous Cell Carcinoma (HNSCC)PET-CT Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 12-5378-CE
Record Dates: First submitted 2014-11-27; First posted 2016-02-10 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck Squamous Cell Carcinoma; Radiation therapy; Head and Neck Cancers
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HNSCC Patients receiving RT (Experimental)
  Interventions: Drug: 18-F FDG

INTERVENTIONS:
Drug: 18-F FDG — All patients enrolled in this study will receive 2 PET Scans: One prior to Radiation, and one during Radiation.

SUMMARY:
The purpose of this study is to see how useful the information provided from Positron Emission Tomography (PET) scans can be in the actual planning and delivery of radiation treatment to patients who have head and neck cancers. Patients participating in this study, will have (in addition to their routine tests) a PET scan before and during their radiation treatment. Following the intervention, patients will be followed as per standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Non-nasopharynx head and neck mucosal squamous cell carcinoma
* Radiologically evident gross disease
* Radiotherapy alone for curative intent
* Age equal to or more than 18 years old
* To be eligible for the second study PET-CT scan: FDG avid tumour (or minimum SUV of 2.5) on the first study PET-CT scan

Exclusion Criteria:

* Nasopharynx cancer
* H&N SCC skin
* Distant metastases (already known or if found on baseline CT-thorax)
* Prior malignancy within the last 5 years (exclude non-H&N SCC, BCC skin)
* Prior chemotherapy within the last 5 years or concurrent chemotherapy/EGFR inhibitors
* Prior head and neck radiotherapy
* Inability to lie supine for study duration
* Pregnancy
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-10; Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Measure rate constant of 18F-FDG uptake in tumour and normal tissue with dynamic PET scanning before radiotherapy. | ~ 2 years

SECONDARY OUTCOMES:
Measure rate constant of 18F-FDG uptake in tumour and inflammatory tissue with dynamic PET scanning during radiotherapy . | ~ 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John J Kim, MD, Principal Investigator — The Princess Margaret Cancer Foundation
Locations (1):
- University Health Network, Princess Margaret Cancer Center, Toronto, Ontario, Canada